CLINICAL TRIAL: NCT00866255
Title: Continuous Measurement of Intratracheal Pressure in Mechanically Ventilated Infants
Brief Title: Continuous Measurement of Intratracheal Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Dr. med. Daniel Steinmann, University Medical Center Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 237/06
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2009-03

CONDITIONS: Endotracheal Pressure
Keywords: endotracheal tube; endotracheal pressure; airway pressure; pressure drop; calculation; continuous calculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: endotracheal tube pressure measurement probe — The endotracheal tube pressure measurement probe is inserted into the endotracheal tube prior to intubation for measurement of tracheal pressure at the tip of the endotracheal tube.

SUMMARY:
Continuous measurement of intratracheal pressure in mechanically ventilated infants using a fibreoptic pressure transducer in the endotracheal tube (ETT). Based on the findings, tracheal pressure can continuously be monitored in the presence of pediatric ETTs by combining ETT coefficients and the flow and airway pressure continuously measured at the proximal end of the ETT.

ELIGIBILITY:
Inclusion Criteria:

* Children < 10 Years
* volume-controlled ventilation

Exclusion Criteria:

* refusal of written informed consent
* severe pulmonary diseases

Ages: 1 Day to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
tracheal pressure | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Freiburg, Freiburg im Breisgau, Germany

REFERENCES:
- [Background] Guttmann J, Kessler V, Mols G, Hentschel R, Haberthur C, Geiger K. Continuous calculation of intratracheal pressure in the presence of pediatric endotracheal tubes. Crit Care Med. 2000 Apr;28(4):1018-26. doi: 10.1097/00003246-200004000-00018. PMID 10809276
- [Background] Guttmann J, Eberhard L, Fabry B, Bertschmann W, Wolff G. Continuous calculation of intratracheal pressure in tracheally intubated patients. Anesthesiology. 1993 Sep;79(3):503-13. doi: 10.1097/00000542-199309000-00014. PMID 8363076
- [Derived] Spaeth J, Steinmann D, Kaltofen H, Guttmann J, Schumann S. The pressure drop across the endotracheal tube in mechanically ventilated pediatric patients. Paediatr Anaesth. 2015 Apr;25(4):413-20. doi: 10.1111/pan.12595. Epub 2014 Dec 10. PMID 25491944